CLINICAL TRIAL: NCT03278925
Title: A Phase I Single-arm, Multicenter Pilot Study Aimed at Validating γ-OHPdG as a Biomarker and Testing the Effects of Polyphenon E on Its Levels in Patients With Cirrhosis
Brief Title: Defined Green Tea Catechin Extract in Preventing Liver Cancer in Participants With Cirrhosis
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2017-01557; NCI-2017-01557 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN-2012-00035; NCI 2016-08-02 (Other: Northwestern University); NWU2016-08-02 (Other: DCP); N01CN00035 (NIH); P30CA060553 (NIH)
Record Dates: First submitted 2017-09-11; First posted 2017-09-12 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (defined green tea catechin extract) (Experimental): Participants receive defined green tea catechin extract PO QD or BID for 24 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo ultrasound, CT, or MRI at screening and on study, undergo collection of blood samples on study, and may undergo biopsy at screening and on study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Defined Green Tea Catechin Extract; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Other: Pharmacological Study; Other: Questionnaire Administration; Procedure: Ultrasound

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Defined Green Tea Catechin Extract — Given PO
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Pharmacological Study — Correlative studies
Other: Questionnaire Administration — Ancillary studies
Procedure: Ultrasound — Undergo ultrasound

SUMMARY:
This phase I trial studies the side effects and best dose of defined green tea catechin extract and to see how well it works in preventing liver cancer in participants with cirrhosis. Higher levels of the molecule gamma-OHPdG may be found in participants with cirrhosis, which may mean a higher risk of the development of liver cancer. Defined green tea catechin extract may work better to lower levels of gamma-OHPdG and prevent the development of liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish maximum tolerated dose (MTD) and to collect safety data of defined green tea catechin extract (Polyphenon E/epigallocatechin gallate [EGCG]) treatment in participants with cirrhosis.

II. To determine the effects of Polyphenon E/EGCG treatment on the suppression of gamma-hydroxy-1,N(2)-propanodeoxyguanosine (gamma-OHPdG) levels in cirrhotic liver.

SECONDARY OBJECTIVES:

I. To collect Polyphenon E/EGCG pharmacokinetic data in participants with cirrhosis.

II. To determine the effects of Polyphenon E/EGCG treatment on the suppression of gamma-hydroxy-1,N(2)-propanodeoxyguanosine (gamma-OHPdG) levels in cirrhotic liver by liquid chromatography-mass spectrometry (LC-MS) assay from baseline to post-treatment.

III. To estimate the fraction of participants with liver cirrhosis that have high levels of gamma-OHPdG.

EXPLORATORY OBJECTIVES:

I. To assess the effects of Polyphenon E/EGCG on the grade of cirrhosis as measured by FibroScan (registered trademark) and Fibrosis-4 (FIB-4) score.

II. To develop a LC-MS and/or enzyme-linked immunosorbent assay (ELISA)-based method for detecting urinary and blood gamma-OHPdG, to correlate with liver gamma-OHPdG levels.

III. To evaluate any hepatocellular carcinoma (HCC) development during the treatment.

OUTLINE: This is a dose-escalation study.

Participants receive defined green tea catechin extract orally (PO) once daily (QD) or twice daily (BID) for 24 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo ultrasound, computed tomography (CT), or magnetic resonance imaging (MRI) at screening and on study, undergo collection of blood samples on study, and may undergo biopsy at screening and on study.

After completion of study intervention, participants are followed up at 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a clinical diagnosis of cirrhosis based on the investigators evaluation, confirmed by ANY ONE of the three following methods to define cirrhosis:

  * Established cirrhosis on liver biopsy (Meta-analysis of Histological Data in Viral Hepatitis [METAVIR] F4);
  * Ultrasound, CT or MRI findings consistent with cirrhosis; nodular appearing liver with or without evidence of portal hypertension
  * Transient elastography (FibroScan) with a result > 12.5 kPa Etiology of cirrhosis will not be considered in determining inclusion in the study
* Participant is able and willing to comply with study procedures, and signed and dated informed consent is obtained
* Participant agrees to consume no more than 2 cups of green tea per day and refrain from taking supplements or foods labeled as containing green tea
* Participant must be aged >= 18 years. Because no dosing or adverse event (AE) data are currently available on the use of Polyphenon E in participants < 18 years of age, children are excluded from this study but will be eligible for future pediatric trials, if applicable
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Platelets >= 75,000 / uL
* Hemoglobin >= 8 g/dL
* Serum creatinine OR measured or calculated creatinine clearance within normal institutional limits; glomerular filtration rate (GFR) can also be used in place of creatinine or creatinine clearance (CrCl) within normal institutional limits as adjusted for age and sex
* Serum direct bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 X upper normal level (UNL)
* Albumin >= 3.0 mg/dL
* International normalized ratio (INR) =< 1.3
* Ascites absent
* Encephalopathy absent
* Only participants found to express high levels (immunohistochemistry [IHC] score 3 and above) of gamma-OHPdG (gamma-OHPdG-high HCC) in baseline or archival liver biopsy will be registered to receive Polyphenon E treatment
* Participant is able to undergo radiographic evaluation with ultrasound, CT, or MRI
* The effects of Polyphenon E on the developing human fetus at the recommended therapeutic dose are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence); contraception must be used prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately; female participants of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication (if a urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required)

Exclusion Criteria:

* Participant has confirmed HCC by ultrasound/CT/MRI; participants who have previously had HCC but have been treated and have been recurrence free for 5 years are eligible
* Participant has or has had other cancer(s) within 3 years of study; however, in situ breast, in situ cervical, and basal cell/squamous cell skin cancers are allowed; participant with active, other cancer that requires systemic therapy will be excluded from this study; participant with early stage cancer that requires local therapy, such as cervical ablation for early stage cervical cancer, are allowed to be registered in the study and are allowed to receive local therapy
* Inability to swallow capsules
* Participant has a known diagnosis of mental incapacitation that may affect their ability to consent and be compliant with the protocol
* Participant has ever experienced one or more hepatic decompensation events or a history of decompensated liver disease as listed below:

  * Clinical ascites
  * Variceal bleeding documented by endoscopy
  * Spontaneous bacterial peritonitis documented by positive culture
  * Hepatic encephalopathy
  * Hepatorenal syndrome (type 1 or 2)
  * Porto-pulmonary hypertension
  * Hepato-pulmonary hypertension
  * Any liver-related event which led to a hospitalization or a grade 4 event
* Participant has an underlying predisposition to gastrointestinal (GI) or rectal bleeding are considered ineligible for study participation
* History of allergic reactions attributed to compounds of similar chemical composition to Polyphenon E (or green tea); note that participants who are unable to tolerate intravenous contrast for CT scans should have MRIs or ultrasounds during the study instead of CT scans
* Participant is receiving any other investigational agents
* Participants have taken supplements or foods that are labelled as containing green tea for 8 weeks before start of treatment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; hepatitis b virus (HBV) and hepatitis C virus (HCV) infections are allowed
* Green tea has been consumed by humans for thousands of years and teratogenic or abortifacient effects have not been reported; however, subjects in this study will take high doses of Polyphenon E; the teratogenic or abortifacient effects of high dose Polyphenon E is unknown; therefore pregnant women are excluded from this study; because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother with Polyphenon E, breastfeeding should be discontinued if the mother is treated with this study agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of Polyphenon E | Up to 4 weeks
  Will be defined as the dose at which =< 1 subjects out of 6 experiences a grade 3 or higher toxicity based on Common Terminology Criteria for Adverse Events criteria.
Change in gamma-hydroxy-1,N(2)-propanodeoxyguanosine (gamma-OHPdG) expression in cirrhotic liver | Baseline up to 24 weeks
  Will be assessed by immunohistochemistry. Will use a nonparametric Wilcoxon test to compare the post-pre differences to zero.

SECONDARY OUTCOMES:
Fraction of patients with liver cirrhosis that have high levels of gamma-OHPdG | Up to 24 weeks
  Will use descriptive statistics.
Change in gamma-OHPdG | Baseline up to 24 weeks
  Descriptive statistics (mean, range) will be used to summarize this continuous outcome by dose level. A nonparametric trend test will be used to examine whether there is a trend for greater reduction in gamma-OHPdG as the dose level increases.
Polyphenon E pharmacokinetic data in blood and urine in patients with cirrhosis | Prior to and at 1.5, 3.5, and 8.5 hours after the first dose of Polyphenon E on day 1
  Clearance of Polyphenon E will be compared among cirrhotic liver patients in this study and results from this population will be compared with non-cirrhotic historical control participants.

OTHER OUTCOMES:
Grade of cirrhosis | Up to 24 weeks
  Will be assessed by FibroScan and Fibrosis-4 score.
Liquid chromatography-mass spectrometry (LC-MS) and/or enzyme-linked immunosorbent assay (ELISA)-based method for detecting gamma-OHPdG | Up to 24 weeks
  The research urine samples at screen 2 and research blood samples collected at visit 1, visit 2, and Visit 3 will be used to develop a non-invasive LC-MS and/or ELISA-based method to quantify gamma-OHPdG in urine and blood samples of collected from trial participants. Descriptive statistics (n; minimum; maximum; mean; median; standard deviation for continuous variables; and n, frequency for categorical variables) will be used to summarize participants demographics. Participants safety data will be tabulated according to the symptom and grade. Estimates will be presented with their 95% confidence intervals.
Incidence of hepatocellular carcinoma | At baseline and 24 weeks
  Evaluated using ultrasound/computed tomography/magnetic resonance imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Aiwu R He, Principal Investigator — Northwestern University
Locations (2):
- MedStar Georgetown University Hospital, Washington D.C., District of Columbia, United States
- University of Puerto Rico, San Juan, Puerto Rico

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT03278925/Prot_SAP_000.pdf